CLINICAL TRIAL: NCT05576350
Title: Evaluation of a Combined Motivational Interviewing and Ecological Momentary Intervention to Reduce Risky Alcohol Use Among Individuals Vulnerable to HIV/AIDS
Brief Title: TRAC-ER Intervention to Reduce Risky Alcohol Use and HIV Risk
Acronym: TRAC-ER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Yale University (Other)
Responsible Party: Principal Investigator, Carolyn Lauckner, Associate Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 79109; 1R01AA030487-01 (NIH)
Record Dates: First submitted 2022-09-29; First posted 2022-10-12 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Risk Behavior; Alcohol Use Disorder; HIV Infections
Keywords: motivational interviewing; behavior; ecological momentary intervention; EMI; TRAC; mobile; GPS
MeSH Terms: conditions — Risk-Taking; Alcoholism; HIV Infections; Behavior | interventions — Ethanol; Economics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SAM-Only Comparison Group (Experimental): Participants in this group will engage only in smartphone-based alcohol monitoring.
  Interventions: Behavioral: Smartphone Based Alcohol Monitoring (SAM)
- TRAC plus SAM (Experimental): Participants in this group will receive the Tracking and Reducing Alcohol Consumption (TRAC) intervention and smartphone-based alcohol monitoring.
  Interventions: Behavioral: Smartphone Based Alcohol Monitoring (SAM); Behavioral: Tracking and Reducing Alcohol Consumption (TRAC)
- TRAC-ER plus SAM (Experimental): Participants in this group will receive the Tracking and Reducing Alcohol Consumption (TRAC) intervention combined with GPS-based ecological momentary interventions (EMI) and smartphone-based alcohol monitoring.
  Interventions: Behavioral: Smartphone Based Alcohol Monitoring (SAM); Behavioral: Tracking and Reducing Alcohol Consumption (TRAC); Behavioral: TRAC-ER

INTERVENTIONS:
Behavioral: Smartphone Based Alcohol Monitoring (SAM) — Smartphone-based alcohol monitoring (SAM) using mobile breathalyzers and surveys.
Behavioral: Tracking and Reducing Alcohol Consumption (TRAC) — The TRAC intervention focuses on increasing motivation and building skills for avoiding triggers and managing situations that encourage drinking. It requires four 30-minute sessions with a counselor using videoconferencing and mobile phones. In addition to receiving the four sessions of intervention content, participants will complete smartphone-based self-monitoring of alcohol consumption, which will be discussed during intervention sessions.
  Arms: TRAC plus SAM; TRAC-ER plus SAM
Behavioral: TRAC-ER — Ecological momentary interventions (EMI) use phones to deliver messages to reduce alcohol use and related risk behaviors during or prior to drinking events. GPS tracking can determine when individuals visit places they have previously reported drinking or triggers to drink and then EMI messages can be delivered upon arrival to prevent risky alcohol use.
  Arms: TRAC-ER plus SAM

SUMMARY:
Ecological momentary interventions (EMI), which use phones to deliver messages to reduce alcohol use and related risk behaviors during or prior to drinking events, can help to address triggers in real-time. GPS tracking can determine when individuals visit places they have previously reported drinking or triggers to drink and then EMI messages can be delivered upon arrival to prevent risky alcohol use. A mobile app has been developed that uses GPS tracking to determine when individuals visit "risky" places and then delivers a survey asking what behaviors they engaged in while at the location.

The goal of the proposed study is to use this app to enhance the Tracking and Reducing Alcohol Consumption (TRAC) intervention by delivering messages that encourage participants to employ strategies discussed during TRAC sessions when arriving at risky places. When they leave these places, they will complete a survey and breathalyzer reading in order to collect event-level self-report and biological data on alcohol use and HIV risk. If their breathalyzer result indicates alcohol use, they will receive harm reduction messaging. It is expected that combining TRAC with EMI ("TRAC-ER") will increase effectiveness by reinforcing topics discussed during these sessions, providing in-the-moment messaging to address triggers, and collecting real-time alcohol use data.

DETAILED DESCRIPTION:
For this study, the investigators will enhance an existing mHealth intervention (TRAC) to reduce alcohol use among young adults at risk for HIV by combining the intervention with an app which delivers EMI messages in real-time. Upon enrollment, participants will be randomized into one of 3 arms: TRAC-ER (EMI messaging, TRAC intervention, and smartphone-based alcohol monitoring), TRAC (TRAC intervention and smartphone-based alcohol monitoring), or a comparison group (smartphone-based alcohol monitoring only).

Participants will be recruited from Kentucky and Connecticut through community-based recruitment and health clinics.

Preliminary data used for this study were collected from a study (PI: Lauckner, K01AA02530) testing the TRAC intervention with people living with HIV/AIDS, which has shown promising preliminary results, with high feasibility, acceptability, and encouraging preliminary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* is between the ages of 18-35 at the start of the study
* owns a smartphone
* has not been diagnosed with HIV
* screens positively for at-risk alcohol use (score of 4 or higher on the AUDIT-C, OR report engaging in binge drinking at least once over the past 12 months).
* meets criteria for pre-exposure prophylaxis (PrEP) OR is identified as being at high risk for HIV (i.e., reports history of using PrEP/PEP, reports unprotected sex, etc.)

Exclusion Criteria:

* do not speak English
* are actively detoxifying from substances and need medical supervision
* a score of 20 or greater on the Alcohol Use Disorders Identification Test

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 405 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of drinking days | Measured daily for 30 day periods during months 1, 2, 3, 6, and 9
  Number of days in which alcohol was consumed based on breathalyzer readings greater than 0.00

SECONDARY OUTCOMES:
Number of binge drinking episodes | Measured daily for 30 day periods during months 1, 2, 3, 6, and 9
  Number of binge drinking episodes (occasions when participants had 5+ drinks based on self-reported number of drinks)
Number of drinks/drinking day | Measured daily for 30 day periods during months 1, 2, 3, 6, and 9
  3 items: alcohol consumed (yes or no), number of drinks, and time spent drinking

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Lauckner, PhD, Principal Investigator — University of Kentucky; Trace Kershaw, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - University of Kentucky, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lauckner C, Takenaka BP, Sesenu F, Brown JS, Kirklewski SJ, Nicholson E, Haney K, Adatorwovor R, Boyd DT, Fallin-Bennett K, Restar AJ, Kershaw T. Combined Motivational Interviewing and Ecological Momentary Intervention to Reduce Hazardous Alcohol Use Among Sexual Minority Cisgender Men and Transgender Individuals: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Apr 5;13:e55166. doi: 10.2196/55166. PMID 38578673